CLINICAL TRIAL: NCT05992454
Title: An Evaluation of Manual Ventilation Practices of Professional Firefighters During Cardiopulmonary Resuscitation.
Brief Title: Ventilation in Cardiac Arrest Resuscitation Study
Acronym: VECARS
Status: Completed | Type: Observational
Sponsor: French Defence Health Service (Other Government)
Collaborators: Fire Brigade Of Paris Emergency Medicine Dept (Other)
Responsible Party: Principal Investigator, Daniel Jost, Physician heading the scientific section, Fire Brigade Of Paris Emergency Medicine Dept
Other Study IDs: 2022-A02771-42
Record Dates: First submitted 2023-07-06; First posted 2023-08-15 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Heart Arrest, Out-Of-Hospital; CardioPulmonary Resuscitation; Basic Cardiac Life Support
Keywords: heart arrest; cardiopulmonary resuscitation; bag-valve-mask; rescuers
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: EOLIFE — Measurement of ventilatory parameters during manual ventilation by professional rescuers during out-of-hospital cardiac arrest

SUMMARY:
Out-of-hospital cardiac arrest (OHCA) is a major public health problem, with around 40,000 victims each year in France. Their survival rate remains dramatically low, at less than 10%.

In the event of pre-hospital cardiac arrest, rescuers perform resuscitation techniques using equipment for which they have been trained. They perform cardiopulmonary resuscitation (CPR) by alternating 30 chest compressions with 2 insufflations (30/2) with a manual insufflator bag.

In basic life supports, insufflations should result in chest rise, but guidelines do not specify a precise volume.

Recently, medical devices have been developed that enable precise measurement of ventilatory volumes. In simulation, these devices show hyperventilation in volume and frequency in mannequins. But no clinical study has analyzed insufflator bag ventilation maneuvers in real-life situations on pre-hospital cardiac arrest patients.

The aim of this study is to analyze ventilation parameters in current practice in relation to standards, and the factors influencing the quality of ventilation maneuvers.

ELIGIBILITY:
Inclusion Criteria:

* Out of hospital cardiac arrest with CPR performed by the Firefighters
* Age 18 and over
* BLS team on site before arrival of physician staffed ALS means
* CPR ventilation initially provided with Bag-valve- mask
* Measuring device records ventilatory parameters

Exclusion Criteria:

* trauma related OHCA
* airway obstruction during CPR
* OHCA on hanging
* tracheostomized patient
* obstacle to using the Bag-valve-mask
* CPR time less than 2 minutes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Civilian population in hyperurban areas
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2023-05-26 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Tidal volume | up to 20 minutes (end of BLS-CPR)
  Measurement of volume (mL) provided by the BLS Teams [air + oxygen] for each manual insufflation performed by the rescuer

SECONDARY OUTCOMES:
chest rise | up to 20 minutes (end of BLS-CPR)
  concomitant chest rise (YES/NO) during each ventilation procedure
Ventilation rate | up to 20 minutes (end of BLS-CPR)
  Ventilation rate per min. achieved by the rescuer
Insufflation time | up to 20 minutes (end of BLS-CPR)
  Insufflation time (seconds) per ventilation procedure
Face mask leakage | up to 20 minutes (end of BLS-CPR)
  face mask leakage per ventilation procedure
Volume received by the patient | up to 20 minutes (end of BLS-CPR)
  Volume received (mL) by the patient per ventilation procedure
Survival to day 60 after cardiac arrest | up to 60 days
  Survival curve over the first 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Frederic Lemoine, NP, Principal Investigator — Paris Fire Brigade Emergency Dept; Stephane Travers, MD PhD, Study Chair — Paris Fire Brigade Emergency Dept
Locations (1):
- Paris Fire Brigade, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lemoine F, Jost D, Lemoine S, Petermann A, Salome M, Tassart B, Liscia J, Briche F, Bon O, Derkenne C, Frattini B, Travers S; Paris Fire Brigade Cardiac Arrest Task Force (collaborators). Manual bag-valve-mask ventilation during out-of-hospital cardiopulmonary resuscitation: a prospective observational study. Resuscitation. 2025 Dec;217:110895. doi: 10.1016/j.resuscitation.2025.110895. Epub 2025 Nov 12. PMID 41237844